CLINICAL TRIAL: NCT02042755
Title: Pilot Study With a Diffractive Trifocal IOL (POD AY 26P FineVision)
Status: Completed | Type: Observational
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: POD AY 26P FineVision
Record Dates: First submitted 2013-12-20; First posted 2014-01-23 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Bilateral Cataract
Keywords: cataract; IOL; trifocal; FineVision
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: trifocal intraocular lens — Standard cataract surgery
  Other Names: Physiol POD 26P AY FineVision

SUMMARY:
The principal objective of the study is to determine the visual acuity at far, intermediate and near distances tested with optotypes at different distances from the eyes and tested with defocus addition lenses of patients implanted bilaterally with the POD 26P AY FineVision.

Secondary objective will be to test the glare and contrast sensitivity.

DETAILED DESCRIPTION:
This study is a pilot study. As such it will recruit a limited number of patients : 20. Patients recruited will suffer from cataract, have no comorbidity, expressed the desire for spectacle independence and have realistic expectations.

Descriptive statistics will be used to determine the visual acuities at any distance. The occurence of glare and the determination of the contrast sensitivity will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* - Age-related cataract
* Preoperative Corneal astigmatism < 0.75 D
* Age 21 and older
* Visual Acuity > 0.05
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.
* Patient willing multifocal implantation and with realistic expectations.

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome, floppy iris syndrome, corneal pathologies, retinal pathology (diabetic maculopathy, myopic maculopathy, age related macular degeneration...)
* Previous ocular surgery or trauma.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract patients wishing high spectacle independance after the surgery
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 3 months
  At far, near and intermediate distance.

SECONDARY OUTCOMES:
Contrast sensitivity | 3 months
  Assessment of the contrast sensitivity: determination of the visual acuity with low-contrast chart (Pelli Robson standard sight-chart ).

CONTACTS AND LOCATIONS:
Overall Officials: Irit Bahar, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center 49Th Jabotinsky Street, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No